CLINICAL TRIAL: NCT04903041
Title: A Cardiac Registry to Evaluate and Manage the hsTnI Categorical CVD Risk in Subjects Undergoing Preventive Health Checks (PHC).
Status: Suspended | Type: Observational
Why Stopped: Unavailable funding
Sponsor: Jaime Marino (Industry)
Collaborators: Apollo Hospitals Enterprise Limited (Other)
Responsible Party: Sponsor-Investigator, Jaime Marino, Sr Medical Affairs Manager, Abbott Diagnostics Division
Organization: Abbott Diagnostics Division (Industry)
Other Study IDs: ACCR
Record Dates: First submitted 2021-05-12; First posted 2021-05-26 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiovascular disease is the leading cause of mortality globally. In India cardiovascular disease leads to death a decade earlier than in western countries. In the past 20 years awareness and classic risk factors and statins have been the main improvements. However, all these factors have not decreased the cardiovascular disease burden. One reason may be because all of the current assessments for cardiac risk are correlants to disease and none are specific to cardiac myocyte status.

DETAILED DESCRIPTION:
Development of high-sensitivity assays for cardiac troponin I (hs-TnI) has enhanced the ability to detect low circulating levels of cardiac troponins, which are often present in individuals with common cardiac conditions and risk factors who have not manifested clinical cardiovascular disease (CVD). Lowering the detection threshold of troponin assays has expanded the potential use of cardiac troponins from a diagnostic tool in the setting of acute coronary syndrome to a biomarker for risk stratification in individuals without known CVD. Detectable levels of cardiac troponins have been associated with increased incidence of coronary heart disease (CHD), heart failure (HF), and cardiovascular mortality in community-based studies.

Traditional cardiovascular risk prediction does not identify everyone who will develop cardiovascular disease with up to 50% of individuals having none or only one risk factor at the time of diagnosis. Although traditional risk estimations perform moderately well, there remain significant limitations in their use in the prevention of cardiovascular disease especially at an individual level. At an individual level, the clinician not only needs to correctly identify those at increased risk, but also weigh up the importance of each risk factor and determine who needs medical therapy in addition to lifestyle advice Many risk estimation systems in existence are based on a core set of cardiovascular risk factors and based on participants either selected randomly from the general population or those attending their general practitioner. All these risk scoring systems show a good level of discrimination, for cardiovascular events, with the area under the receiving operator curve ranging from 0.73 to 0.82. However, adopting these risk scoring systems to guide current clinical practice has limitations. First, most of these scoring systems, except QRISK1 and QRISK2 have been developed from old prospective cohorts with participants recruited in the 1980's and 1990's Second, applying risk estimation scores to regions with different rates of baseline rates of cardiovascular disease will lead to either under- or over-estimation of risk: a result of mis-calibration. Third, the value of incorporating new risk factors including biomarkers such as high-sensitivity C reactive protein has been disappointing in improving discrimination, with age and sex alone contributing to 0.70 of the area under the receiver operating curve statistic. None of these risk estimation scores, to date, incorporate a direct measure of cardiac injury such as cardiac troponin and its potential role in guiding primary prevention in a contemporaneous population remains uncertain.

ELIGIBILITY:
Inclusion Criteria:

1. All men and women above the age of 18 years
2. Lipid profiles ordered
3. HbA1c ordered
4. Creatinine ordered

Exclusion Criteria:

1. Non-consenting subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects undergoing health checks at Apollo Group of hospitals in Hyderabad, Chennai, Bangalore, Mumbai, Kolkata and New Delhi.
Sampling Method: Non-Probability Sample
Enrollment: 300000 (Estimated)
Dates: Start 2019-09-12 (Actual); Primary Completion 2029-09-12 (Estimated); Study Completion 2030-09-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the hsTnI categorical CVD risk model with the Apollo Healthcare system in subjects attending the Preventive Health Checkups. | Through study completion, an average of 1 year
  Number of individuals classified as high, moderate, low risk based on the pre-defined cut-offs of high-sensitivity troponin I.

SECONDARY OUTCOMES:
Implementation of recommendation for the low, moderate and high risk in subjects and monitoring the outcome in the cardiac registry database. | Through study completion, an average of 1 year
  Number of individuals that follows the cardiovascular risk stratification algorithm: lifestyle consultation, treatment of underlying conditions such as hypertension, diabetes, hyperlipidemia as well as ECG, stress test echocardiography recommendations and number of individuals experiencing the adverse cardiovascular outcomes per cardiovascular risk category.

OTHER OUTCOMES:
Optimize the use of hsTnI risk categories by clinicians | Through study completion, an average of 1 year
  Estimate the longitudinal changes of the number of clinicians that recommend the following based on the cardiovascular risk stratification algorithm: lifestyle consultation, treatment of underlying conditions such as hypertension, diabetes, hyperlipidemia as well as ECG, stress test and echocardiography recommendations.

CONTACTS AND LOCATIONS:
Overall Officials: Pratap C Reddy, MD, Principal Investigator — Apollo Hopsitals; Hari Prasad, MD, Principal Investigator — Apollo Hospitals Enterprise Limited; Abraham Oomman, MD, Principal Investigator — Apollo Hospitals Enterprise Limited; Padma Madala, MD, Principal Investigator — Apollo Hospitals Enterprise Limited; Jaganathan Sickan, MD, Principal Investigator — Abbott; Agim Beshiri, MD, Principal Investigator — Abbott
Locations (6):
- India (6):
  - Apollo Hospitals, Bangalore
  - Apollo Hospitals, Chennai
  - Apollo Hospitals, Hyderabad
  - Apollo Hospitals, Kolkata
  - Apollo Hospitals, Mumbai
  - Apollo Hospitals, New Delhi

IPD SHARING:
Plan to Share IPD: No
No plan to share with other researchers

REFERENCES:
- [Background] Lankeit M, Jimenez D, Kostrubiec M, Dellas C, Hasenfuss G, Pruszczyk P, Konstantinides S. Predictive value of the high-sensitivity troponin T assay and the simplified Pulmonary Embolism Severity Index in hemodynamically stable patients with acute pulmonary embolism: a prospective validation study. Circulation. 2011 Dec 13;124(24):2716-24. doi: 10.1161/CIRCULATIONAHA.111.051177. Epub 2011 Nov 14. PMID 22082681
- [Background] Xue Y, Clopton P, Peacock WF, Maisel AS. Serial changes in high-sensitive troponin I predict outcome in patients with decompensated heart failure. Eur J Heart Fail. 2011 Jan;13(1):37-42. doi: 10.1093/eurjhf/hfq210. Epub 2010 Dec 13. PMID 21149316
- [Background] Rosjo H, Varpula M, Hagve TA, Karlsson S, Ruokonen E, Pettila V, Omland T; FINNSEPSIS Study Group. Circulating high sensitivity troponin T in severe sepsis and septic shock: distribution, associated factors, and relation to outcome. Intensive Care Med. 2011 Jan;37(1):77-85. doi: 10.1007/s00134-010-2051-x. Epub 2010 Oct 12. PMID 20938765
- [Background] Afonso L, Bandaru H, Rathod A, Badheka A, Ali Kizilbash M, Zmily H, Jacobsen G, Chattahi J, Mohamad T, Koneru J, Flack J, Weaver WD. Prevalence, determinants, and clinical significance of cardiac troponin-I elevation in individuals admitted for a hypertensive emergency. J Clin Hypertens (Greenwich). 2011 Aug;13(8):551-6. doi: 10.1111/j.1751-7176.2011.00476.x. Epub 2011 Jun 27. PMID 21806764
- [Background] Hoiseth AD, Neukamm A, Karlsson BD, Omland T, Brekke PH, Soyseth V. Elevated high-sensitivity cardiac troponin T is associated with increased mortality after acute exacerbation of chronic obstructive pulmonary disease. Thorax. 2011 Sep;66(9):775-81. doi: 10.1136/thx.2010.153122. Epub 2011 Jun 8. PMID 21653926
- [Background] de Lemos JA, Drazner MH, Omland T, Ayers CR, Khera A, Rohatgi A, Hashim I, Berry JD, Das SR, Morrow DA, McGuire DK. Association of troponin T detected with a highly sensitive assay and cardiac structure and mortality risk in the general population. JAMA. 2010 Dec 8;304(22):2503-12. doi: 10.1001/jama.2010.1768. PMID 21139111
- [Background] deFilippi CR, de Lemos JA, Christenson RH, Gottdiener JS, Kop WJ, Zhan M, Seliger SL. Association of serial measures of cardiac troponin T using a sensitive assay with incident heart failure and cardiovascular mortality in older adults. JAMA. 2010 Dec 8;304(22):2494-502. doi: 10.1001/jama.2010.1708. Epub 2010 Nov 15. PMID 21078811
- [Background] Meune C, Reichlin T, Irfan A, Schaub N, Twerenbold R, Meissner J, Reiter M, Luthi A, Haaf P, Balmelli C, Drexler B, Winkler K, Hochholzer W, Osswald S, Mueller C. How safe is the outpatient management of patients with acute chest pain and mildly increased cardiac troponin concentrations? Clin Chem. 2012 May;58(5):916-24. doi: 10.1373/clinchem.2011.178053. Epub 2012 Mar 12. PMID 22410086